CLINICAL TRIAL: NCT05766319
Title: The ICU-recover Box, Using Smart Technology for Monitoring Health Status After ICU Admission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Sesmu M. Arbous, MD PhD MSc, dr., Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL81044.058.22
Record Dates: First submitted 2022-11-11; First posted 2023-03-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Critically Ill; ICU Survivor; User Experience
Keywords: E-health; Home monitoring devices; Smartphone-enabled; Health monitoring devices; Smart devices; User experience
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: 10 patients who have been admitted to the ICU, at the Leiden University Medical Centre, and have been discharged to home will be using home monitoring for 3 consecutive months after hospital discharge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving the ICU-recover box containing home monitoring devices (Experimental): Treatment of subjects on the ICU will be state of the art, conform current practice, protocols and guidelines.
  Patients discharged from the ICU will receive an ICU-Recover Box on one of the clinical wards of the LUMC filled with several devices after they have given informed consent. These devices are listed below and are described in further detail in section 6 of this protocol.
  The ICU-Recover Box contains the following devices and tools:
  * Withings BPM Connect
  * Withings Body weight scale
  * Withings ScanWatch, from which the following features will be used:
    * Measurement of SpO2
    * Automatic recording of heart rate
    * Automatic recording of activity (step count)
  Interventions: Device: Withings ScanWatch; Device: Withings BPM Connect; Device: Withings Body

INTERVENTIONS:
Device: Withings ScanWatch — Withings ScanWatch, from which the following features will be used:
  * Measurement of peripheral oxygen saturation (%)
  * Automatic recording of heart rate (beats/min)
  * Automatic recording of activity (step count) (numbers/day)
Device: Withings BPM Connect — Withings BPM connect, from which the following feature will be used:
  o Measurement of non invasive bloodpressure (mmHg)
Device: Withings Body — Withings Body (Scale), from which the following feature will be used:
  o Measurement of body weight (kg)

SUMMARY:
In this pilot study we will study the feasibility of providing and following ICU patients with smart technology for three months after discharge from a general ward of the Leiden University Medical Centre.

DETAILED DESCRIPTION:
Rationale: Smart technology could improve quality of care in patients who have been admitted to the ICU and have been discharged from ICU and hospital, by early diagnosis of complications and early (ambulatory) treatment.

In times of increasing medical care consumption leading to increasing health care costs the investigators have to adopt new ways of acquiring patient-specific knowledge and new ways of delivering care. To obtain this level of insight the investigators need a smart and connected health care system. With the ICU-Recover Box and its smart technology we see new opportunities to improve patient health and to recognise early if escalation of medical care is needed. By intervening early the investigators can reduce costs by reducing health care utilization.

Objectives: The primary objective of the pilot study is to assess the feasibility of the introduction and use of smart technology by persons that have been discharged from the ICU in the three months following hospital discharge. If this pilot study proves to be successful, smart technology will be used in future studies.

Study design: This is a single center cohort study. Study population: The study population consists of 15 patients who have been discharged from the ICU Department to a general ward of the Leiden University Medical Centre.

Intervention: Patients who consent to take part in the study, receive an ICU-Recover Box closely before hospital discharge on the general ward. The ICU-Recover Box will contain a smartphone compatible blood pressure monitor, weight scale, and a watch containing a peripheral oxygen saturation monitor, a pedometer to monitor activity for home monitoring. Never will results of any of the measurements be used for therapy or diagnosis.

Main study parameters/endpoints: The primary endpoint of the study will be the feasibility of providing and following ICU patients with smart technology for three months after discharge from a general ward of the Leiden University Medical Centre.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Patient has been admitted to the ICU of the LUMC for > 48 hours.
* Patient has received mechanical ventilation for > 24 hours.
* Patient masters the English or Dutch language.
* Patient is able and capable to use smart technology at home. (i.e. Wi-Fi available, sufficient comprehension of smart technology).
* Patient can be contacted and informed about the ICU-Recover box on one of the clinical wards of the LUMC.
* Patient is discharged from a ward within the LUMC to home..

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* Patient is < 18 years old.
* Patient is pregnant.
* Patient breastfeeds during the course of the study
* Patient underwent cardiothoracic surgery (as they will receive the Cardiothoracic Box in another study).
* Patient is discharged for palliative care.
* Patient is considered an incapacitated adult.
* Patient is unwilling to sign the informed consent form.
* Patient is discharged to another hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of using home monitoring devices in terms of patient number | three months
  Primary endpoint of this study is the feasibility of providing patients with the ICU-Recover Box after ICU discharge and before hospital discharge, including the collection of measurement/questionnaire data after hospital discharge. This study will be used to identify the issues when implementing such a system. Feasibility is defined as:
  10 post-ICU patients, who gave informed consent and who were discharged from hospital with the ICU-Recover Box, were able to use the devices within its intended use.
Feasibility of using home monitoring devices in terms of data acquisition | three months
  We were able to acquire data from the devices in the ICU-Recover Box.
  * Heart rate ( beats/min ) from the Withings ScanWartch
  * steps/day from the Withings ScanWatch
  * peripheral oxygen saturation (%) from the Withings ScanWatch
  * weight ( kg) from Withings Body
  * Blood pressure ( mmHg) from Withings BPM Connect
Feasibility of using home monitoring devices in terms of data storage | three months
  · We were able to store the acquired data in a safe manner in the datasafe of the LUMC
Feasibility of using home monitoring devices in terms of data analyzability | three to six months
  · We were able to analyse the acquired data (using Python).
Feasibility of using home monitoring devices | six months
  · · > 80 % of the persons that were discharged with an ICU-Recover Box contributed for three months to post-ICU data

SECONDARY OUTCOMES:
Acceptability of home monitoring | three months
  Secondary endpoints are:
  · Users, i.e. post-ICU patients, have been asked, by short interviews, for feedback and suggested a
Improvements of home monitoring | three months
  · By means of PDCA cycli, the lessons learned and feedback will have led to adjustment and improvement of the ICU-Recover Box, from its content and its use to data acquisition and data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sesmu Arbous, MD PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in home monitoring of ICU survivors. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a data transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis. This is subject to individual patient consent.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). This is also subject to individual patient consent. For more information or to submit a request, the principal investigator or a member of the research team can be contacted.